CLINICAL TRIAL: NCT01743911
Title: Phosphodiesterase-5 Inhibitor (Tadalafil) Two Weeks Administration Period Effects in Left Ventricle Diastolic Dysfunction and BNP Levels in Resistant Hypertensive Patients
Brief Title: Tadalafil Effects in Left Ventricle Diastolic Dysfunction in Resistant Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Heitor Moreno Junior, MD, PhD., University of Campinas, Brazil
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE 0044.0.146.000-09; [2009/53430-7] (Other: FAPESP)
Record Dates: First submitted 2012-11-30; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Hypertension
Keywords: Tadalafil; Resistant Hypertension; Left Ventricle Diastolic Dysfunction; Brain natriuretic peptide
MeSH Terms: conditions — Hypertension | interventions — Sugars; Tadalafil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugar pill (Placebo Comparator): Intervention: sugar pill
  Interventions: Other: sugar pill
- tadalafil (Active Comparator): Intervention: tadalafil
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Other: sugar pill — Sugar pills: 20mg orally, once a day for 2 weeks
  Other Names: No brand name.
  Arms: sugar pill
Drug: Tadalafil — Tadalafil pills: 20mg orally, once a day for 2 weeks.
  Other Names: Cialis, Lilly, USA
  Arms: tadalafil

SUMMARY:
Left ventricle diastolic dysfunction (LVDD) is associated with resistant hypertension. In addition, brain natriuretic peptide (BNP) levels are elevated when LVDD is present. It has been shown that phosphodiesterase-5 (PDE5) inhibition improves left ventricle diastolic function in hypertensive rats, despite any difference in blood pressure levels. Also, left ventricle diastolic function enhancement reduces BNP concentration in hypertensive patients. However, it is unknown if these effects exists in humans with resistant hypertension. Therefore, this study was developed to evaluate if the use of a PDE5 inhibitor (tadalafil) for 2 weeks improves LVDD and its effects in BNP levels in resistant hypertensive patients.

DETAILED DESCRIPTION:
Resistant hypertensive patients have a high incidence of left ventricle diastolic dysfunction (LVDD). Lowering blood pressure levels improves diastolic function, however, there is no proved effective treatment specifically for this disease. Studies in hypertensive rats have shown presence of phosphodiesterase-5 in cardiac cells and an improvement in left ventricle diastolic function using a phosphodiesterase-5 (PDE5) inhibitor, the sildenafil. PDE5 has also been demonstrated in human heart cells with cardiac disease. In addition, LVDD is associated with high levels of brain natriuretic peptide (BNP), which reduces with diastolic function improvement. Therefore, it is reasonable to suppose that PDE-5 inhibitor use in humans with LVDD and resistant hypertension could improve diastolic function. Objective: Evaluate the chronic effect of a PDE-5 inhibitor on LVDD and BNP levels in resistant hypertensive patients. Casuistic and methods: 20 resistant hypertensive patients with LVDD types I and II will be evaluated with echocardiography study, ambulatory blood pressure monitoring (ABPM), office blood pressure measurements, endothelial function analysis using the brachial artery flow mediation dilation technique (FMD) and BNP plasma levels. Then, the subjects will receive oral placebo for 2 weeks. After this period, the same exams will be repeated. Two weeks later, the protocol will be performed again to the same 20 patients, using tadalafil (the longest half-life PDE-5 inhibitor) 20mg orally instead of the placebo. Hypothesis: investigators hypothesize that the use of tadalafil will improve left ventricle diastolic function with BNP reduced levels and this effect will be independent of blood pressure decrease or endothelial function improvement.

ELIGIBILITY:
Inclusion Criteria:

* resistant hypertension (according to Resistant Hypertension - American Heart Association Statement - 2008);
* compliance with antihypertensive treatment;
* age >35 years;
* left ventricle diastolic dysfunction types I and II

Exclusion Criteria:

* valvulopathy
* decompensated heart failure
* important cardiac arrhythmias
* nephropathy
* hepatopathy
* autoimmune disease
* tabagism
* decompensated diabetes
* uncontrolled dislipidemia

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricle Diastolic Dysfunction | Baseline and 2 weeks
  Outcome measurement assessed by Echocardiogram before and after a 2-week tadalafil administration period.

SECONDARY OUTCOMES:
Change in endothelial function | baseline and 2 weeks
  Outcome measure assessed by flow-mediated dilation before and after a 2-week tadalafil administration period.
Change in blood pressure levels | Baseline and 2 weeks
  Blood pressure measurements assessed before and after a 2-week tadalafil administration period.
Change in B-type Natriuretic Peptide (BNP-32) levels | Baseline and 2 weeks
  Plasma brain natriuretic peptide (BNP-32)assessed before and after a 2-week tadalafil administration period
Change in cyclic guanosine monophosphate (cGMP) levels | Baseline and 2 weeks
  Cyclic guanosine monophosphate (cGMP) levels assessed before and after a 2-week tadalafil administration period
Change in nitrite levels | Baseline and 2 weeks
  Nitrite levels assessed before and after a 2-week tadalafil administration period.

CONTACTS AND LOCATIONS:
Overall Officials: Heitor Moreno-Junior, MD, PhD, Principal Investigator — Faculty of Medical Sciences - Unicamp
Locations (1):
- Laboratory of Cardiovascular Pharmacology - FCM - Unicamp, Campinas, São Paulo, Brazil